CLINICAL TRIAL: NCT01404312
Title: Phase III Clinical Trial of Ultra-Short-Course Rifapentine/Isoniazid for the Prevention of Active Tuberculosis in HIV-Infected Individuals With Latent Tuberculosis Infection
Brief Title: Brief Rifapentine-Isoniazid Evaluation for TB Prevention (BRIEF TB)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A5279; 10848 (Registry Identifier: DAIDS ES Registry Number); ACTG A5279 (Other: Network)
Record Dates: First submitted 2011-07-26; First posted 2011-07-28 (Estimated); Results first posted 2018-12-06 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2020-12

CONDITIONS: Tuberculosis; HIV Infections
MeSH Terms: conditions — Tuberculosis; HIV Infections | interventions — rifapentine; Isoniazid; Pyridoxine; Vitamin B 6

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RPT plus INH Regimen (Arm A) (Experimental): Participants received RPT (dosage based on their weight), 300 mg of INH, and 25 mg or 50 mg of pyridoxine (vitamin B6) each day during Weeks 1 to 4. During Weeks 5 to 36, participants did not receive any study medications.
  Interventions: Drug: Rifapentine (RPT); Drug: Isoniazid (INH); Dietary Supplement: Pyridoxine (Vitamin B6)
- INH Regimen (Arm B) (Active Comparator): Participants received 300 mg of INH and 25 mg or 50 mg of pyridoxine (vitamin B6) each day during Weeks 1 to 36.
  Interventions: Drug: Isoniazid (INH); Dietary Supplement: Pyridoxine (Vitamin B6)

INTERVENTIONS:
Drug: Rifapentine (RPT) — RPT dosing was be based on participants' weight:
  Participants who weighed 30 kg to less than 35 kg received 300 mg once daily (administered as two 150-mg tablets).
  Participants who weighed 35 kg to less than 45 kg received 450 mg once daily (administered as three 150-mg tablets).
  Participants who weighed greater than 45 kg received 600 mg once daily (administered as four 150-mg tablets).
  Arms: RPT plus INH Regimen (Arm A)
Drug: Isoniazid (INH) — Participants received one 300-mg tablet or three 100-mg tablets of INH once daily.
Dietary Supplement: Pyridoxine (Vitamin B6) — Participants received 25 mg or 50 mg of pyridoxine, based on the current local, national, or international dosing guidelines.
  Participants who received 25 mg of pyridoxine took one 25-mg tablet once daily with INH.
  Participants who received 50 mg of pyridoxine took two 25-mg tablets once daily with INH.

SUMMARY:
HIV-infected people have an increased risk of developing active tuberculosis (TB). At the time the study was designed, the standard course of treatment for TB was 6 to 9 months of isoniazid (INH).This study compared the safety and effectiveness of a 4-week regimen of rifapentine (RPT) plus INH versus a standard 9-month regimen of INH in HIV-infected people who are at risk of developing active TB.

DETAILED DESCRIPTION:
The World Health Organization (WHO) estimated that in 2017 there were 10 million new cases of TB, and 1.6 million people died as a result of TB. Among new TB cases, it is estimated that 920,000 occurred in people who were HIV-coinfected, and 23% of TB deaths were among HIV-coinfected individuals. In Africa, TB is the leading AIDS-related opportunistic infection. Latent TB infection occurs when people are infected with the bacteria that cause TB, but they do not have any symptoms of TB infection. Latent TB can develop into active TB, and HIV-infected people have an increased risk of progressing from latent TB to active TB. INH is a medication that is prescribed for people with latent TB to help prevent active TB from developing. The standard INH treatment regimen is 6 to 9 months; a shorter treatment regimen of 3 months of once-weekly RPT plus INH has proven to be as effective and improved adherence. The purpose of this study was to compare the safety and effectiveness of a 4-week daily regimen of RPT plus INH to a standard 9-month daily INH regimen for TB prevention in HIV-infected individuals.

This study enrolled HIV-infected people who did not have evidence of active TB but who were at high risk of developing active TB. Participants were randomly assigned to receive RPT and INH once a day for 4 weeks or INH once a day for 9 months. All participants received pyridoxine (vitamin B6) with each dose of INH to help prevent possible side effects. Study visits occurred at baseline and Weeks 2, 4, 8, 12, 16, 20, 24, and 36. At select study visits, participants had a physical exam, clinical assessment, blood collection, and a chest radiograph or chest computed tomography (CT) scan (if needed). Some participants had their blood stored for future testing. Follow-up study visits occurred every 12 weeks starting at Week 48 and continued for 3 years after the last participant enrolled.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* Tuberculin skin test (TST) reactivity greater than or equal to 5 mm or a positive interferon gamma release assay (IGRA) at any time prior to study entry, OR living in a high TB burden area. More information on this criterion can be found in the protocol.
* Laboratory values obtained within 30 days prior to study entry:

  1. Absolute neutrophil count (ANC) greater than 750 cells/mm^3
  2. Hemoglobin greater than or equal to 7.4 g/dL
  3. Platelet count greater than or equal to 50,000/mm^3
  4. AST (SGOT) and ALT (SGPT) less than or equal to three times the upper limit of normal (ULN)
  5. Total bilirubin less than or equal to 2.5 times the ULN
* Chest radiograph or chest CT scan without evidence of active tuberculosis, unless one has been performed within 30 days prior to entry
* Female participants of reproductive potential must have a negative serum or urine pregnancy test performed within 7 days prior to study entry. More information on this criterion can be found in the protocol.
* All participants must agree not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, donate sperm, in vitro fertilization) while receiving RPT and for 6 weeks after stopping this drug
* Female participants who are participating in sexual activity that could lead to pregnancy must agree to use one reliable non-hormonal form of contraceptive while receiving RPT and for 6 weeks after stopping this drug. More information on this criterion can be found in the protocol.
* Weight of greater than or equal to 30 kg
* Participant or legal guardian is able and willing to provide informed consent

Exclusion Criteria:

* Treatment for active or latent TB (pulmonary or extrapulmonary) within 2 years prior to study entry or, at screening, presence of any confirmed or probable TB based on criteria listed in the current ACTG Diagnosis Appendix
* History of multi-drug resistant (MDR) or extensively-drug resistant (XDR) TB at any time prior to study entry
* Known exposure to MDR or XDR TB (e.g., household member of a person with MDR or XDR TB) at any time prior to study entry
* Treatment for more than 14 consecutive days with a rifamycin or more than 30 consecutive days with INH at any time during the 2 years prior to enrollment
* For participants taking antiretroviral therapy (ART) at study entry, only approved nucleoside reverse transcriptase inhibitors (NRTIs) with efavirenz (EFV) or nevirapine (NVP) for at least 4 weeks were permitted
* History of liver cirrhosis at any time prior to study entry.
* Evidence of acute hepatitis, such as abdominal pain, jaundice, dark urine, and/or light stools within 90 days prior to study entry
* Diagnosis of porphyria at any time prior to study entry
* Peripheral neuropathy greater than or equal to Grade 2 according to the December 2004 (Clarification, August 2009) Division of AIDS (DAIDS) Toxicity Table, within 90 days prior to study entry
* Known allergy/sensitivity or any hypersensitivity to components of study drugs or their formulation
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Serious illness requiring systemic treatment and/or hospitalization within 30 days prior to study entry
* Breastfeeding

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Actual)
Dates: Start 2012-05-23 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E. Chaisson, MD, Study Chair — Johns Hopkins University; Susan Swindells, MBBS, Study Chair — University of Nebraska
Locations (45):
- United States (21):
  - University of California, UC San Diego CRS- Mother-Child-Adolescent HIV Program, La Jolla, California
  - University of Southern California CRS, Los Angeles, California
  - UCSD Antiviral Research Center CRS, San Diego, California
  - Ucsf Hiv/Aids Crs, San Francisco, California
  - Harbor-UCLA CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Denver Public Health CRS, Denver, Colorado
  - The University of Miami AIDS Clinical Research Unit (ACRU) CRS, Miami, Florida
  - Northwestern University CRS, Chicago, Illinois
  - Boston Medical Center CRS, Boston, Massachusetts
  - Henry Ford Hosp. CRS, Detroit, Michigan
  - Cooper Univ. Hosp. CRS, Camden, New Jersey
  - New Jersey Medical School Clinical Research Center CRS, Newark, New Jersey
  - Nyu Ny Nichd Crs, New York, New York
  - Columbia P&S CRS, New York, New York
  - Bronx-Lebanon Hospital Center NICHD CRS, The Bronx, New York
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Duke University Medical Center CRS, Durham, North Carolina
  - Trinity Health and Wellness Center CRS, Dallas, Texas
  - Houston AIDS Research Team CRS, Houston, Texas
  - University of Washington AIDS CRS, Seattle, Washington
- Botswana (2):
  - Gaborone CRS, Gaborone
  - Molepolole CRS, Gaborone
- Brazil (6):
  - Hospital Nossa Senhora da Conceicao CRS, Porto Alegre, Rio Grande do Sul
  - Univ. of Sao Paulo Brazil NICHD CRS, São Paulo, São Paulo
  - Hospital Federal dos Servidores do Estado NICHD CRS, Rio de Janeiro
  - Instituto de Pesquisa Clinica Evandro Chagas (IPEC) CRS, Rio de Janeiro
  - Hosp. Geral De Nova Igaucu Brazil NICHD CRS, Rio de Janeiro
  - Inst de Infectologia Emilio Ribas Sao Paulo Brazil NICHD CRS, São Paulo
- Haiti (2):
  - Les Centres GHESKIO Clinical Research Site (GHESKIO-INLR) CRS, Port-au-Prince
  - GHESKIO Institute of Infectious Diseases and Reproductive Health (GHESKIO - IMIS) CRS, Port-au-Prince
- Kenya (3):
  - Kisumu Crs, Kisumu, Nyanza
  - Kenya Medical Research Institute/Walter Reed Project Clinical Research Center (KEMRI/WRP) CRS, Kericho, Rift Valley
  - Moi University Clinical Research Center (MUCRC) CRS, Eldoret
- Malawi (2):
  - Malawi CRS, Lilongwe, Central Region
  - Blantyre CRS, Blantyre
- Peru (2):
  - Barranco CRS, Lima
  - San Miguel CRS, Lima
- South Africa (3):
  - Soweto ACTG CRS, Johannesburg, Gauteng
  - Wits Helen Joseph Hospital CRS (Wits HJH CRS), Johannesburg, Gauteng
  - Durban International Clinical Research Site CRS, Durban, KwaZulu-Natal
- Thailand (3):
  - Thai Red Cross AIDS Research Centre (TRC-ARC) CRS, Bangkok
  - Chiang Mai University HIV Treatment (CMU HIV Treatment) CRS, Chiang Mai
  - Chonburi Hosp. CRS, Chon Buri
- Parirenyatwa CRS, Harare, Zimbabwe

REFERENCES:
- [Background] Golub JE, Pronyk P, Mohapi L, Thsabangu N, Moshabela M, Struthers H, Gray GE, McIntyre JA, Chaisson RE, Martinson NA. Isoniazid preventive therapy, HAART and tuberculosis risk in HIV-infected adults in South Africa: a prospective cohort. AIDS. 2009 Mar 13;23(5):631-6. doi: 10.1097/QAD.0b013e328327964f. PMID 19525621
- [Background] Zhang T, Zhang M, Rosenthal IM, Grosset JH, Nuermberger EL. Short-course therapy with daily rifapentine in a murine model of latent tuberculosis infection. Am J Respir Crit Care Med. 2009 Dec 1;180(11):1151-7. doi: 10.1164/rccm.200905-0795OC. Epub 2009 Sep 3. PMID 19729664
- [Derived] Pham MM, Podany AT, Mwelase N, Supparatpinyo K, Mohapi L, Gupta A, Samaneka W, Omoz-Oarhe A, Langat D, Benson CA, Chaisson RE, Swindells S, Fletcher CV. Population Pharmacokinetic Modeling and Simulation of Rifapentine Supports Concomitant Antiretroviral Therapy with Efavirenz and Non-Weight Based Dosing. Antimicrob Agents Chemother. 2022 Sep 20;66(9):e0238521. doi: 10.1128/aac.02385-21. Epub 2022 Aug 9. PMID 35943252
- [Derived] Haas DW, Podany AT, Bao Y, Swindells S, Chaisson RE, Mwelase N, Supparatpinyo K, Mohapi L, Gupta A, Benson CA, Baker P, Fletcher CV. Pharmacogenetic interactions of rifapentine plus isoniazid with efavirenz or nevirapine. Pharmacogenet Genomics. 2021 Jan;31(1):17-27. doi: 10.1097/FPC.0000000000000417. PMID 32815870
- [Derived] Miyahara S, Ramchandani R, Kim S, Evans SR, Gupta A, Swindells S, Chaisson RE, Montepiedra G. Applying a Risk-benefit Analysis to Outcomes in Tuberculosis Clinical Trials. Clin Infect Dis. 2020 Feb 3;70(4):698-703. doi: 10.1093/cid/ciz784. PMID 31414121
- [Derived] Swindells S, Ramchandani R, Gupta A, Benson CA, Leon-Cruz J, Mwelase N, Jean Juste MA, Lama JR, Valencia J, Omoz-Oarhe A, Supparatpinyo K, Masheto G, Mohapi L, da Silva Escada RO, Mawlana S, Banda P, Severe P, Hakim J, Kanyama C, Langat D, Moran L, Andersen J, Fletcher CV, Nuermberger E, Chaisson RE; BRIEF TB/A5279 Study Team. One Month of Rifapentine plus Isoniazid to Prevent HIV-Related Tuberculosis. N Engl J Med. 2019 Mar 14;380(11):1001-1011. doi: 10.1056/NEJMoa1806808. PMID 30865794
- [Derived] Podany AT, Bao Y, Swindells S, Chaisson RE, Andersen JW, Mwelase T, Supparatpinyo K, Mohapi L, Gupta A, Benson CA, Kim P, Fletcher CV; AIDS Clinical Trials Group A5279 Study Team. Efavirenz Pharmacokinetics and Pharmacodynamics in HIV-Infected Persons Receiving Rifapentine and Isoniazid for Tuberculosis Prevention. Clin Infect Dis. 2015 Oct 15;61(8):1322-7. doi: 10.1093/cid/civ464. Epub 2015 Jun 16. PMID 26082504
- See also: DIVISION OF AIDS TABLE FOR GRADING THE SEVERITY OF ADULT AND PEDIATRIC ADVERSE EVENTS VERSION 1.0, DECEMBER, 2004; CLARIFICATION AUGUST 2009 — https://rsc.niaid.nih.gov/sites/default/files/table-for-grading-severity-of-adult-pediatric-adverse-events.pdf
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS — http://rsc.tech-res.com/docs/default-source/safety/manual_for_expedited_reporting_aes_to_daids_v2.pdf?sfvrsn=12

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-five Clinical Research sites across 10 countries participated in the study. The first participant was randomized on May 23, 2012. Accrual closed on November 12, 2014 with 3,000 participants enrolled in the study.
Pre-assignment Details: Randomization was 1:1, and stratified by CD4 count (< 100, 100-250, and > 250 cells/mm^3), and antiretroviral therapy status (receiving antiretroviral therapy or not receiving antiretroviral therapy at enrollment).
Groups:
- RPT Plus INH Regimen (Arm A): Participants received RPT (dosage based on their weight), 300 mg of INH, and 25 mg or 50 mg of pyridoxine (vitamin B6) each day during Weeks 1 to 4. During Weeks 5 to 36, participants did not receive any study medications.
  Rifapentine (RPT): RPT dosing was based on participants' weight:
  Participants who weighed 30 kg to less than 35 kg received 300 mg once daily (administered as two 150-mg tablets).
  Participants who weighed 35 kg to less than 45 kg received 450 mg once daily (administered as three 150-mg tablets).
  Participants who weighed greater than 45 kg will receive 600 mg once daily (administered as four 150-mg tablets).
  Isoniazid (INH): Participants received one 300-mg tablet or three 100-mg tablets of INH once daily.
  Pyridoxine (Vitamin B6): Participants received 25 mg or 50 mg of pyridoxine, based on the current local, national, or international dosing guidelines.
  Participants receiving 25 mg of pyridoxine took one 25-mg tablet once daily
- INH Regimen (Arm B): Participants received 300 mg of INH and 25 mg or 50 mg of pyridoxine (vitamin B6) each day during Weeks 1 to 36.
  Isoniazid (INH): Participants received one 300-mg tablet or three 100-mg tablets of INH once daily.
  Pyridoxine (Vitamin B6): Participants received 25 mg or 50 mg of pyridoxine, based on the current local, national, or international dosing guidelines.
  Participants receiving 25 mg of pyridoxine took one 25-mg tablet once daily with INH.
  Participants receiving 50 mg of pyridoxine took two 25-mg tablets once daily with INH.
Period: Overall Study
Arm/Group | RPT Plus INH Regimen (Arm A) | INH Regimen (Arm B)
Started | 1496 | 1504
Completed | 1198 | 1193
Not Completed | 298 | 311
Not completed — Death | 21 | 27
Not completed — Withdrawal by Subject | 15 | 18
Not completed — Participant Unable to get to clinic | 93 | 103
Not completed — Lost to Follow-up | 115 | 111
Not completed — Site closed | 22 | 21
Not completed — Participant not willing to adhere to req | 31 | 29
Not completed — Severe debilitation, unable to continue | 1 | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | RPT Plus INH Regimen (Arm A) | INH Regimen (Arm B) | Total
Number analyzed (Participants) | 1496 | 1504 | 3000
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (10.3) | 35.6 (10.3) | 35.7 (10.3)
Age, Customized [Count of Participants; unit: Participants]
  Age at Entry: <=20 years | 77 | 70 | 147
  Age at Entry: >20, <=30 years | 421 | 455 | 876
  Age at Entry: >30, <=40 years | 523 | 514 | 1037
  Age at Entry: >40, <=50 years | 342 | 331 | 673
  Age at Entry: >50 years | 133 | 134 | 267
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 802 | 812 | 1614
  Male | 694 | 692 | 1386
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White Non-Hispanic | 16 | 12 | 28
  Race/Ethnicity: Black Non-Hispanic | 992 | 991 | 1983
  Race/Ethnicity: Hispanic (Regardless of Race) | 361 | 369 | 730
  Race/Ethnicity: Asian, Pacific Islander | 122 | 128 | 250
  Race/Ethnicity: Not Reported | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  Haiti | 198 | 198 | 396
  United States | 45 | 46 | 91
  Malawi | 106 | 108 | 214
  Botswana | 210 | 212 | 422
  Brazil | 102 | 98 | 200
  South Africa | 307 | 309 | 616
  Zimbabwe | 56 | 58 | 114
  Kenya | 93 | 94 | 187
  Thailand | 121 | 124 | 245
  Peru | 258 | 257 | 515
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.6 (5.2) | 24.5 (5.3) | 24.5 (5.2)
IV Drug Use [Count of Participants; unit: Participants]
  Never | 1489 | 1497 | 2986
  Currently | 2 | 1 | 3
  Previously | 5 | 6 | 11
Prior Tuberculosis History [Count of Participants; unit: Participants]
  Yes | 82 | 89 | 171
  No | 1414 | 1415 | 2829
Screening CD4 counts [Count of Participants; unit: Participants]
  <100 cells/mm^3 | 37 | 37 | 74
  >=100,<=250 cells/mm^3 | 160 | 165 | 325
  >250 cells/mm^3 | 1299 | 1302 | 2601
Antiretroviral Therapy (ART) at Entry [Count of Participants; unit: Participants]
  Efavirenz-based | 650 | 649 | 1299
  Nevirapine-based | 97 | 100 | 197
  Neither Efavirenz nor Nevirapine-based | 3 | 6 | 9
  Not on ART | 746 | 749 | 1495
HIV-1 RNA Viral load among participants on ART at entry [Count of Participants; unit: Participants] — Undetectable defined as HIV-1 RNA < 40 copies/mL Population: Measured only in those participants who were taking antiretroviral therapy at entry.
  Participants
    number analyzed (Participants) | 750 | 755 | 1505
    Detectable | 154 | 143 | 297
    Undetectable | 569 | 586 | 1155
    Not Reported | 27 | 26 | 53

OUTCOME MEASURES:

1. Primary Outcome: Incidence of First Diagnosis of Active Tuberculosis, Death Related to Tuberculosis, or Death From Unknown Cause
Description: Incidence rate (events per 100 person-years) was estimated, and 95.1% confidence interval used to account for interim analysis of primary efficacy outcome.
Time Frame: From entry to occurrence of event, up to end of follow-up 3 years after last participant enrolled (median follow-up time: 3.3 years)
Population: All participants who started study treatment.
Measure: Number (95.1% Confidence Interval); unit: Events per 100 person-years
Arm/Group | RPT Plus INH Regimen (Arm A) | INH Regimen (Arm B)
Number analyzed (Participants) | 1488 | 1498
Events per 100 person-years | 0.6506 [0.4242 to 0.8770] | 0.6736 [0.4428 to 0.9045]
Statistical Analysis 1: Comparison: RPT Plus INH Regimen (Arm A) vs INH Regimen (Arm B); Mantel-Haenszel method used for estimating standardized incidence rate in each arm and incidence rate difference; Test type: Non-Inferiority — Non-inferiority margin: 1.25 events per 100 person-years. Sample size determination was based on the assumption of a primary endpoint rate of 2.0/100 person-years, with a one-sided 0.025 alpha level, and targeting at least 90% power. This required a sample size of approximately 2500. The sample size was adjusted upwards to account for loss to follow-up, interim monitoring, and to allow for subgroup analyses with reasonable power; Incidence Rate Difference = -0.0231, 95.1% CI 2-sided [-0.346 to 0.300] — Estimate given as Incidence rate in Arm A - Incidence Rate in Arm B (negative favors Arm A). Incidence rate units: Events per 100 person-years

2. Secondary Outcome: Number of Participants With Occurrence of One or More Serious Adverse Events (SAEs) Versus no SAEs
Description: Occurrence of any SAE that meets the ICH definition of an SAE
Time Frame: as for outcome 1
Population: All participants who started study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | RPT Plus INH Regimen (Arm A) | INH Regimen (Arm B)
Number analyzed (Participants) | 1488 | 1498
Participants
  No SAE occurred | 1405 | 1390
  At least one SAE occurred | 83 | 108
Statistical Analysis 1: Comparison: RPT Plus INH Regimen (Arm A) vs INH Regimen (Arm B); Comparison of the proportion of participants with any SAE occurrence between arms A and B. H0: Proportion of participants with SAE in Arm A = Proportion of participants with SAE in Arm B; Test type: Superiority; p = 0.073, Fisher Exact — Not adjusted for multiple comparisons; Risk Difference (RD) = -0.016, 95% CI 2-sided [-0.035 to 0.002] — Estimate given as: Proportion Arm A - Proportion Arm B

3. Secondary Outcome: Number of Participants With a Targeted Adverse Event
Description: Targeted adverse events include each new grade 3 or 4 laboratory value or sign or symptom that is at least one grade increase from baseline for the following: nausea and vomiting; cutaneous; drug-associated fever; elevated aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]), alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]), or bilirubin; and peripheral neuropathy
Time Frame: as for outcome 1
Population: All participants who started study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | RPT Plus INH Regimen (Arm A) | INH Regimen (Arm B)
Number analyzed (Participants) | 1488 | 1498
Participants
  No Targeted Safety Event | 1445 | 1446
  Occurrence of Targeted Safety Event | 43 | 52
Statistical Analysis 1: Comparison: RPT Plus INH Regimen (Arm A) vs INH Regimen (Arm B); Comparison of the proportion of participants with any targeted adverse event occurrence between arms A and B. H0: Proportion of participants with a targeted adverse event in Arm A = Proportion of participants with a targeted adverse event in Arm B; Test type: Superiority; p = 0.405, Fisher Exact — Not adjusted for multiple comparisons; Risk Difference (RD) = -.0058, 95% CI 2-sided [-0.019 to 0.007] — Estimate given as: Proportion Arm A - Proportion Arm B

4. Secondary Outcome: Number of Participants in Each Category of Ordered Categorical Variable Indicating Most Stringent Level of Study Drug Management Due to Toxicity That Was Required Over the Treatment Period
Description: Ordered categories include:
  1. Premature permanent treatment discontinuation
  2. Treatment hold for more than 7 consecutive days
  3. None of the above
Time Frame: From entry to end of treatment (up to 8 weeks for Arm A; up to 54 weeks for Arm B)
Population: All participants who started study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | RPT Plus INH Regimen (Arm A) | INH Regimen (Arm B)
Number analyzed (Participants) | 1488 | 1498
Participants
  Premature permanent treatment discontinuation | 16 | 25
  Treatment held for more than 7 days | 11 | 31
  None of the above | 1461 | 1442
Statistical Analysis 1: Comparison: RPT Plus INH Regimen (Arm A) vs INH Regimen (Arm B); Odds ratio of being in higher category estimated from proportional odds model H0: Odds ratio of being in higher category for Arm A vs Arm B = 1; Test type: Superiority; Odds Ratio (OR) = 2.093, 95% CI 2-sided [1.315 to 3.332] — Estimate given as: Odds of being in higher category (more stringent management due to toxicity) for Arm B compared with arm A Not adjusted for multiple comparisons

5. Secondary Outcome: Cumulative Incidence of Death From Any Cause
Description: Data table estimates for percentage who died by each time point were estimated using Kaplan-Meier at 1, 2, 3, and 4 years post-entry.
Time Frame: as for outcome 1
Population: All Participants who started study treatment
Measure: Number; unit: events per 100 participants
Arm/Group | RPT Plus INH Regimen (Arm A) | INH Regimen (Arm B)
Number analyzed (Participants) | 1488 | 1498
events per 100 participants
  1 year post-entry | 0.35 | 0.63
  2 years post-entry | 0.49 | 1.15
  3 years post-entry | 1.05 | 1.62
  4 years post-entry | 2.00 | 2.29
Statistical Analysis 1: Comparison: RPT Plus INH Regimen (Arm A) vs INH Regimen (Arm B); H0: Survival curve Arm A = Survival curve Arm B; Test type: Superiority; p = 0.3078, Log Rank — Not adjusted for multiple comparisons

6. Secondary Outcome: Cumulative Incidence of Death Due to a Non-TB Event
Description: Cumulative incidence function estimated nonparametrically, treating TB-related deaths as competing risks.
Time Frame: as for outcome 1
Population: All participants who started study treatment
Measure: Number; unit: events per 100 participants
Arm/Group | RPT Plus INH Regimen (Arm A) | INH Regimen (Arm B)
Number analyzed (Participants) | 1488 | 1498
events per 100 participants
  Cumulative incidence by 1 year post-randomization | 0.3 | 0.5
  Cumulative incidence by 2 years post-randomization | 0.4 | 1.0
  Cumulative incidence by 3 years post-randomization | 0.9 | 1.5
  Cumulative incidence by 4 years post-randomization | 1.6 | 2.0
Statistical Analysis 1: Comparison: RPT Plus INH Regimen (Arm A) vs INH Regimen (Arm B); Competing risk analysis using the Fine-Gray model, treating TB-related deaths as competing risks, and other deaths including deaths of unknown cause as the event of interest. H0: Hazard Ratio for Arm A vs Arm B = 1; Test type: Superiority; p = 0.2802, Hazard Ratio — Not adjusted for multiple comparisons; Hazard Ratio (HR) = 1.396, 95% CI 2-sided [0.762 to 2.559] — Hazard ratio given as: Arm B hazard / Arm A hazard, i.e. HR > 1 favors arm A

7. Secondary Outcome: Number of Participants With Antibiotic Resistance Among Mycobacterium Tuberculosis (MTB) Isolates in Participants Who Develop Active Tuberculosis
Description: Among MTB-diagnosed participants who underwent drug-susceptibility testing, the number who had any resistance to a particular drug.
Time Frame: After TB diagnosis
Population: Participants with a culture-confirmed TB diagnosis who underwent drug susceptibility testing
Measure: Count of Participants; unit: Participants
Arm/Group | RPT Plus INH Regimen (Arm A) | INH Regimen (Arm B)
Number analyzed (Participants) | 15 | 12
Participants
  Rifampin: Developed Resistance | 1 | 1
  Rifampin: Did not Develop Resistance | 14 | 11
  Isoniazid: number analyzed (Participants) | 14 | 12
  Isoniazid: Developed Resistance | 2 | 1
  Isoniazid: Did not Develop Resistance | 12 | 11
  Ethambutol: number analyzed (Participants) | 7 | 8
  Ethambutol: Developed Resistance | 0 | 1
  Ethambutol: Did not Develop Resistance | 7 | 7
  Pyrazinamide: number analyzed (Participants) | 6 | 6
  Pyrazinamide: Developed Resistance | 0 | 0
  Pyrazinamide: Did not Develop Resistance | 6 | 6

8. Secondary Outcome: Efavirenz (EFV) Plasma Concentrations in Arm A
Description: Mean and standard deviation.
  Week 16 samples have not yet been analyzed because the metabolite assay is being validated, and requires submission for approval by the Clinical Pharmacology Quality Assurance Program. Analysis of week 16 samples are anticipated to be available in September 2019.
Time Frame: Measured at Weeks 0, 2, 4, and 16
Population: Only measured in the first 90 participants randomized to Arm A who entered the study taking EFV and who meet dose timing criteria; and, under Version 2.0 of the protocol, at Weeks 0, 2, 4, and 16 in the first 30 participants randomized to Arm A who enter the study taking EFV and who meet dose timing criteria.
Measure: Mean (Standard Deviation); unit: nanograms per mL
Arm/Group | RPT Plus INH Regimen (Arm A)
Number analyzed (Participants) | 111
nanograms per mL
  Week 0: number analyzed (Participants) | 99
  Week 0 | 3787 (4922)
  Week 2: number analyzed (Participants) | 110
  Week 2 | 3870 (7011)
  Week 4: number analyzed (Participants) | 87
  Week 4 | 4082 (4916)
  Week 16: number analyzed (Participants) | 0

9. Secondary Outcome: Nevirapine (NVP) Plasma Concentrations in Arm A
Description: Mean and standard deviation
Time Frame: Measured at Weeks 0, 2, and 4
Population: Only measured in the first 90 participants randomized to Arm A who enter the study taking NVP and who meet dose timing criteria. For weeks 0, 2, 4, some samples were missing or contaminated.
Measure: Mean (Standard Deviation); unit: nanograms per mL
Arm/Group | RPT Plus INH Regimen (Arm A)
Number analyzed (Participants) | 90
nanograms per mL
  Week0: number analyzed (Participants) | 88
  Week0 | 7573 (3789)
  Week 2: number analyzed (Participants) | 88
  Week 2 | 6234 (4283)
  Week 4 | 5797 (3963)

10. Secondary Outcome: EFV Plasma Concentrations in Arm B
Description: For Version 2.0 of the protocol only, measured in the first 90 participants randomized to Arm B who enter the study taking EFV and who meet dose timing criteria.
  Outcome measure was not assessed because no participants enrolled under version 2.0 of the protocol were on Efavirenz at study entry.
Time Frame: Measured at weeks 0, 2 and 4
Population: Outcome measure was not assessed because no participants enrolled under version 2.0 of the protocol were on Efavirenz at study entry.
Arm/Group | INH Regimen (Arm B)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From entry to end of follow-up 3 years after last participant enrolled (median follow-up time: 3.3 years)
Description: At entry, all diagnoses, signs/symptoms, and laboratory values of all grades that occurred 30 days before entry were collected; post-entry, all diagnoses regardless of grade, signs/symptoms of grade 3 or higher, laboratory values grade 3 or higher, and all events that led to a change in treatment were collected.
  The DAIDS AE Grading Table (V1.0) and Expedited AE Manual (V2.0) were used.
Groups:
- RPT Plus INH Regimen (Arm A): Participants received RPT (dosage based on their weight), 300 mg of INH, and 25 mg or 50 mg of pyridoxine (vitamin B6) each day during Weeks 1 to 4. During Weeks 5 to 36, participants did not receive any study medications.
  Rifapentine (RPT): RPT dosing was based on participants' weight:
  Participants who weighed 30 kg to less than 35 kg received 300 mg once daily (administered as two 150-mg tablets).
  Participants who weighed 35 kg to less than 45 kg received 450 mg once daily (administered as three 150-mg tablets).
  Participants who weighed greater than 45 kg received 600 mg once daily (administered as four 150-mg tablets).
- INH Regimen (Arm B): Pyridoxine (Vitamin B6): Participants received 25 mg or 50 mg of pyridoxine, based on the current local, national, or international dosing guidelines.
  Participants receiving 25 mg of pyridoxine took one 25-mg tablet once daily
  INH Regimen (Arm B) Participants received 300 mg of INH and 25 mg or 50 mg of pyridoxine (vitamin B6) each day during Weeks 1 to 36.
  Isoniazid (INH): Participants received one 300-mg tablet or three 100-mg tablets of INH once daily.
  Pyridoxine (Vitamin B6): Participants received 25 mg or 50 mg of pyridoxine, based on the current local, national, or international dosing guidelines.
  Participants receiving 25 mg of pyridoxine took one 25-mg tablet once daily with INH.
  Participants receiving 50 mg of pyridoxine took two 25-mg tablets once daily with INH.
Arm/Group | RPT Plus INH Regimen (Arm A) | INH Regimen (Arm B)
All-Cause Mortality (participants affected / at risk) | 21/1496 | 27/1504
Serious Adverse Events (participants affected / at risk) | 40/1496 | 68/1504
Other Adverse Events (participants affected / at risk) | 1051/1496 | 1042/1504
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RPT Plus INH Regimen (Arm A) (N=1496) | INH Regimen (Arm B) (N=1504)
Anaemia (Blood and lymphatic system disorders) | 2 | 3
Neutropenia (Blood and lymphatic system disorders) | 5 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Bundle branch block right (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Death (General disorders) | 1 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 2
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 2 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1
Abscess jaw (Infections and infestations) | 0 | 1
Acute hepatitis B (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Bone tuberculosis (Infections and infestations) | 0 | 1
Breast abscess (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Dengue haemorrhagic fever (Infections and infestations) | 0 | 1
Disseminated tuberculosis (Infections and infestations) | 0 | 2
Encephalitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
HIV infection (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2
Retroviral infection (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Typhus (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Stab wound (Injury, poisoning and procedural complications) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 7
Transaminases increased (Investigations) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebellar ischaemia (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Idiopathic intracranial hypertension (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 4
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Superior sagittal sinus thrombosis (Nervous system disorders) | 1 | 0
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 2 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RPT Plus INH Regimen (Arm A) (N=1496) | INH Regimen (Arm B) (N=1504)
Abdominal pain (Gastrointestinal disorders) | 81 | 83
Diarrhoea (Gastrointestinal disorders) | 101 | 108
Pyrexia (General disorders) | 198 | 187
Nasopharyngitis (Infections and infestations) | 93 | 84
Pharyngitis (Infections and infestations) | 89 | 57
Tonsillitis (Infections and infestations) | 79 | 65
Upper respiratory tract infection (Infections and infestations) | 118 | 117
Alanine aminotransferase increased (Investigations) | 102 | 121
Aspartate aminotransferase increased (Investigations) | 94 | 118
Blood albumin decreased (Investigations) | 97 | 125
Blood alkaline phosphatase increased (Investigations) | 99 | 99
Blood pressure increased (Investigations) | 83 | 63
Blood sodium decreased (Investigations) | 219 | 200
Blood sodium increased (Investigations) | 87 | 107
Haemoglobin decreased (Investigations) | 112 | 120
Neutrophil count decreased (Investigations) | 189 | 146
Weight decreased (Investigations) | 74 | 105
Headache (Nervous system disorders) | 155 | 149
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 93 | 102
Cough (Respiratory, thoracic and mediastinal disorders) | 254 | 238
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 125 | 123
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 202 | 166
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 122 | 130
Hypertension (Vascular disorders) | 95 | 75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights

DOCUMENTS (2):
  • Study Protocol (2014-08-28): https://cdn.clinicaltrials.gov/large-docs/12/NCT01404312/Prot_001.pdf
  • Statistical Analysis Plan (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/12/NCT01404312/SAP_000.pdf